CLINICAL TRIAL: NCT06928688
Title: Assessment of Glycemic Index for Dried Saskatoon Berries and Powder in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS26810 (B2025:012)
Record Dates: First submitted 2025-03-31; First posted 2025-04-15 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers (HV)
Keywords: Postprandial glucose; Glycemic index; blood glucose

STUDY DESIGN:
Intervention Model Description: Volunteers will receive SB powder, whole dried SB fruit or glucose drink with matching carbohydrate as control with 1 week interval between any two tests.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SB powder (Experimental): Volunteers drink 25 g of SB powder (25g carbohydrate equivalent) with 250ml water (consumption within 10 minutes)
  Interventions: Dietary Supplement: Saskatoon berry powder
- Dried whole SB fruit (Experimental): Volunteers intake Dried whole SB fruit (25g carbohydrate equivalent) within 20 minutes. Participants have option to choose intake one or both SB products. One week interval is required between the interventions.
  Interventions: Dietary Supplement: Saskatoon berry powder

INTERVENTIONS:
Dietary Supplement: Saskatoon berry powder — After oral intake of SB powder, dried whole SB fruit or glucose drink, finger tip blood glucose will be measured 15, 30, 45, 60, 90 and 120 minutes after the consumption.
  Other Names: Dried whole Saskatoon berry; Glucose drink as control

SUMMARY:
The glycemic index (GI) ranks carbohydrate-containing foods based on their effect on postprandial blood glucose levels. Foods or food products with lower GI values (55 or less) are absorbed more slowly, gradually increasing blood glucose and insulin levels. Fruits are believed to have a lower GI, making them potentially beneficial for individuals seeking to manage blood sugar levels. Previous studies from our and other groups suggest that Saskatoon berry (SB) is a potential functional food for glucose management. The glycemic index (GI) of dried SB powder and whole fruit remains undetermined, limiting our ability to make precise dietary recommendations. This study aims to evaluate the GI in both whole fruit and powder forms of SB. The determination of GI on SB products allows us to provide evidence-based guidance for healthcare providers when recommending SB as a functional food for glucose control.

DETAILED DESCRIPTION:
I. Research Objective: This study aims to evaluate the GI of Saskatoon berry powder and whole fruit in healthy individuals.

II. Methodology:

Study Design

* Type: Randomized, open-label study.
* Duration: Approximately 4 weeks for each participant.
* Setting: Clinical nutrition laboratory.

Participant Recruitment:

Following approval from the University of Manitoba Research Ethics Board, we will distribute recruitment materials across the university campus. Interested individuals may contact the research coordinator to express interest in participation.

Target enrollment: 10-20 participants

Eligibility Requirements:

* Individuals in good health (males and females)
* Between 18 and 74 years of age
* Body Mass Index (BMI) within the range of 18.5-29.9 kg/m²
* Free from diabetes, hyperlipidemia, and hypertension
* Must not be taking medications for diabetes, cholesterol, or blood pressure management.

Required Resources

* Saskatoon berry powder (Prairie Berry Inc.)
* Whole Saskatoon berries (Prairie Berry Inc.)
* Control substance: 25g glucose drink
* Glucose monitoring instruments
* Water (250ml) for powder administration Protocol Overview Visit #1: Initial Session: Research consent The research coordinator will conduct informed consent procedures at an agreed-upon location.
* Initial Assessment:

  * Blood pressure measurement
  * Heart rate monitoring
  * Anthropometric measurements Visit #2: Primary Testing Session
* Preparation Guidelines:

  * Fasting period: 10-14 hours overnight
  * Session start: 9:00 AM
* Testing Protocol:

The participant will receive either Saskatoon berry powder (25g carbohydrate equivalent) with 250ml of water (consumption within 10 minutes), or whole Saskatoon berries (25g carbohydrate equivalent, consumption within 20 minutes) or glucose drink (25 g carbohydrate, consumption with in 10 min).

Blood glucose monitoring schedule:

Initial reading (0 min) 15 minutes post-consumption 30 minutes post-consumption 45 minutes post-consumption 60 minutes post-consumption 90 minutes post-consumption 120 minutes post-consumption Visit #3: Reference Food Assessment Participants will undergo an identical protocol with oral glucose drink (25g carbohydrate equivalent) 2-7 days following the initial assessment.

Important: A minimum 48-hour washout period is required between each test (control or berry preparation).

Analytical Methods The glycemic index will be determined through analysis of blood glucose area under curve (AUC), following established protocols (Brouns et al., 2005).

* GI will be calculated as the ratio of the incremental AUC (iAUC) for SB to the iAUC for glucose drink, multiplied by 100.
* Data will be presented as mean ± standard deviation.
* Paired t-tests or equivalent non-parametric tests will be used to compare iAUC between SB and glucose drink.
* A p-value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Individuals in good health (males and females)
* Between 18 and 74 years of age
* Signed informed consent

Exclusion Criteria:

* Body Mass Index (BMI) >= 30 kg/m²
* Diabetes, hyperlipidemia, and hypertension
* Taking medications for diabetes, cholesterol, or blood pressure

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Glycemic index | 15-120 minutes after consumption dietary supplement
  Glyemic index after the consumption of SB powder or dried whole SB compared to glucose drink

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brouns F, Bjorck I, Frayn KN, Gibbs AL, Lang V, Slama G, Wolever TM. Glycaemic index methodology. Nutr Res Rev. 2005 Jun;18(1):145-71. doi: 10.1079/NRR2005100. PMID 19079901
- [Result] Zhao R, Khafipour E, Sepehri S, Huang F, Beta T, Shen GX. Impact of Saskatoon berry powder on insulin resistance and relationship with intestinal microbiota in high fat-high sucrose diet-induced obese mice. J Nutr Biochem. 2019 Jul;69:130-138. doi: 10.1016/j.jnutbio.2019.03.023. Epub 2019 Apr 9. PMID 31078906